CLINICAL TRIAL: NCT04081597
Title: A Safety, Tolerability, and Pharmacokinetic Study of Single Ascending Doses of STAR-101 in Healthy Subjects
Brief Title: A Study of Single Ascending Doses of STAR-101 in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in Clinical Strategy
Sponsor: Acanthas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ACANTHAS-P1-101
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAR-101 (Experimental): Doses in two of three crossover periods
  Interventions: Drug: Star-101
- Placebo (Placebo Comparator): Matching placebo in one of three periods
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Star-101 — Administered orally
  Arms: STAR-101
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The study will include a single ascending dose approach to evaluate the safety, tolerability, and pharmacokinetic properties of STAR-101 after a single oral administration in healthy participants

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants who are not vasectomized for at least 6 months and having a female partner of childbearing potential (childbearing potential females are defined as women that are neither post-menopausal nor surgically sterile) must agree to use a reliable method of birth control

  1. Simultaneous use of a male condom and, for the female partner, hormonal contraceptives (used since at least 4 weeks) or intra-uterine contraceptive device(placed since at least 4 weeks) or abstain from sexual intercourse from start of study drug dosing until 90 days after dosing with study drug
  2. Simultaneous use of a male condom and, for the female partner, a diaphragm or cervical cap with intravaginally applied spermicide from start of study drug dosing until 90 days after dosing with study drug
  3. Male participants (including vasectomized males) with a pregnant partner must agree to use a condom from start of study drug dosing until 90 days after dosing with study drug
  4. No contraception is required for a vasectomized male, provided his vasectomy was performed 6 months or more prior to screening and his female partner is not pregnant, and for a male participant with a female partner of non-childbearing potential.
  5. A male who was vasectomized less than 6 months prior to screening must follow the same restrictions as a non-vasectomized male
  6. Males participants must not donate sperm at any time from start of study drug dosing until 90 days after study drug dosing
* Healthy female participants must be nonpregnant and not lactating. Female participants of childbearing potential with a non-sterile male partner (sterile male partners are defined as men vasectomized since at least 6 months) must be willing and able to practice effective contraception from the period described below and for at least 30 days after the study completion. For this study, acceptable contraception includes:

  1. Simultaneous use of intrauterine contraceptive device, without hormone release system, placed at least 4 weeks prior to study drug dosing, and cond om for the male partner
  2. Simultaneous use of diaphragm or cervical cap with intravaginally applied spermicide and male condom for the male partner, started at least 21 days prior to study drug dosing
  3. Sexual abstinence if this is usual and preferred lifestyle choice of participant
* Have a body mass index of greater than or equal to (≥18.5) and less than <30.0 kilogram - meter squared (kg/m2) and body weight ≥50.0 kilograms (kg) for males and ≥45.0 kg for females
* Have given informed consent prior to any study specific- procedures.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow Clinical Research Unit (CRU) specific- study procedures.
* Have clinical laboratory test results within normal reference range for the population or Investigator site, or results with acceptable deviations that are judged not clinically significant by the Investigator

Exclusion Criteria:

* Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to study drug dosing, administration of a biological product in context of a clinical research study within 90 days prior to study drug dosing, or currently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have previously completed or withdrawn from this study or any other study investigating STAR-101
* Have a clinically significant history or presence of medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric, immunological, gastrointestinal, renal, metabolic or neurological disease, convulsions, or any clinically significant laboratory abnormality that, in the judgment of the investigator, indicate a medical problem that would preclude study participation
* Have an abnormality in the 12-lead ECG that, in the opinion of the Investigator, increases the risks associated with participating in the study. In addition, participants with the following findings will be excluded:

  1. Confirmed Frederica's corrected QT (QTcF) interval greater than ( >) 450 msec (milliseconds)
  2. Personal or family history (in a first degree relative) of QT prolongation.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies, hepatitis C and/or positive hepatitis C antibody, or hepatitis B and/or positive hepatitis B surface antigen
* Have donated plasma within 7 days prior to study drug dosing or have donated or lost blood from to 50 (milliliter) mL to 499 mL within 30 days, or more than 499 mL within 56 days prior to study drug dosing
* Are unwilling to stop alcohol and caffeinated beverage consumption for the restriction periods stated
* Use of tobacco or nicotine products within 3 months prior
* Have a history of significant alcohol abuse within 1 year prior or an average weekly alcohol intake that exceeds 14 units per week (1 unit = 12 ounces (oz) or 360 mL of beer; 5oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Have an abnormal blood pressure (supine) defined as diastolic blood pressure >90 or <50 (millimeters of mercury (mmHg) and/or systolic blood pressure >140 or <90 mmHg and/or heart rate>100 bpm or <50 (beats per minute) bpm
* Have following abnormal laboratory results

  1. Alanine transaminase (ALT) or aspartate transaminase (AST) >1.5x upper limit of normal (ULN)
  2. Hemoglobin, white blood cell count, platelets, c-reactive protein, or glucose outside or the normal range
  3. Creatinine above the ULN.
* Participants with a history of drug abuse, considered clinically significant, within 1 year prior to screening or use of soft drugs(such as marijuana) within 3 months prior, or hard drugs (such as cocaine, phencyclidine, crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior, or who test positive for drugs of abuse
* Clinically significant illness or surgery within 4 weeks of study drug dosing
* History of significant allergic reaction or hypersensitivity to any drug
* Positive pregnancy test
* Use of medications for the timeframes specified below, with the exception of medications exempted on a case-by-case basis because they are judged unlikely to affect the pharmacokinetic profile of the study drug or participant safely (for example (e.g.), topical drug products without significant systemic absorption):

  1. Prescription medications within 14 days prior to study drug dosing
  2. Over-the-counter products and natural health products (including herbal remedies such as St. John's wort, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to study drug dosing, with the exception of occasional use of acetaminophen (up to 2 grams (g) daily)
  3. Depot injection or implant of any drug within 3 months prior to study drug dosing
  4. Any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to dosing
* Any reason which, in the opinion of the investigator, would prevent the participant from participating in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Serious Adverse Events (SAEs) | Baseline to approximate 70 days
  A summary of SAEs and other non-serious adverse events (AEs) will be reported in the Adverse Events module
Number of participants with other (non-serious) adverse events | Baseline to approximate 70 days
  A summary of SAEs and other non-serious adverse events (AEs) will be reported in the Adverse Events module

SECONDARY OUTCOMES:
Area under the drug concentration time curve (AUC0 to t-last) | Predose up to 144 hours post dose
  AUC from time zero to last measurable concentration
Area under the drug concentration time curve (AUC0-24) | Predose up to 24 hours postdose
  AUC from time zero to 24 hours
Area under the drug concentration time curve (AUC0-inf) | Predose up to 144 hours post dose
  AUC from time zero to infinity
Maximum observed drug concentration (Cmax) | Predose up to 144 hours post dose
  Cmax of STAR-101
Time to reach Cmax (Tmax) | Predose up to 144 hours post dose
  Tmax of STAR-101
Change in QTc interval | Predose up to 144 hours post dose
  QTc interval

CONTACTS AND LOCATIONS:
Overall Officials: Acanthas Pharma, Study Director — Acanthas Pharma